CLINICAL TRIAL: NCT00216658
Title: Open Label Study to Confirm Effectiveness, Safety and Pharmacokinetics of Fentanyl Transdermal Matrix Patch, in Japanese Patients With Cancer Pain Who Have Had a Minimum Amount of Morphine Therapy, Such as Equal to Less Than 45 mg/Day of Oral Morphine or Oxycodone Equal to Less Than 30 mg/Day.
Brief Title: Phase II Clinical Trial of Fentanyl Transdermal Matrix Patch, in the Management of Cancer Pain- Assessment of Effectiveness, Safety and Pharmacokinetics -
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004876
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Pain, Intractable
Keywords: Fentanyl; Cancer pain; Japanese patients
MeSH Terms: conditions — Pain, Intractable; Cancer Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The purpose of this study is to verify the effectiveness, safety and pharmacokinetics of fentanyl transdermal matrix patches containing either 12.5 mcg/hr, 25 mcg/hr, or 50 mcg/hr in Japanese patients with cancer pain who have been switched from minimum amount of existing morphine preparations, such as equivalent to less than 45 mg/day of oral morphine, or oral oxycodone preparations equivalent to less than 30 mg/day.

DETAILED DESCRIPTION:
Fentanyl transdermal matrix patch is a narcotic analgesic agent. Compared with the existing reservoir-type Durotep® Patch, it is not liable to leakage of drug solution and does not contain alcohol, which becomes a cause of skin irritation. Also this new formulation becomes available of smaller one of 12.5 mcg/hr while the smallest Durotep® Patch is 25 mcg/hr. This clinical trial was planned to assess effectiveness, safety and pharmacokinetics of fentanyl transdermal matrix patch at an initial transdermal dose of 12.5 mcg in Japanese cancer patients with pain receiving morphine preparations equivalent to less than 45 mg/day of oral morphine (less than 30 mg for suppository, less than 15 mg for injection), oral oxycodone preparations equivalent to less than 30 mg/day, or fentanyl citrate injectable solution equivalent to less than 0.3 mg/day. After pre-treatment period for one to three days for evaluating the eligibility of the patients for the study, patients will use 3 patches for 10 days. Starting from the first day of treatment with 12.5 mcg/hr patch, fentanyl will be applied to the chest, the upper arm or other appropriate site, which will be replaced with a new patch every three days (ca. 72 hr). Total treatment duration is ten days, and dose adjustment can be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer pain receiving any of the following treatments constantly for at least 3days before the treatment period :(1)Morphine preparations equivalent to less than 45 mg/day of oral morphine (or less than 30 mg/day of suppositories, or less than 15 mg/day of injectable preparations), (2)oral oxycodone preparations equivalent to less than 30 mg/day, (3)Fentanyl citrate injectable solution equivalent to less than 0.3 mg/day
* Patients with a pain intensity of less than or equal to 34 mm on the 100 mm Visual Analogue Scale (VAS)
* Patients with an established diagnosis of cancer of any type who have been notified of the disease
* Patients may be hospitalized during application of the initial transdermal dose of fentanyl transdermal matrix patch (patients may be ambulatory after the initial patch has been replaced with the second dose)

Exclusion Criteria:

* Patients with respiratory dysfunction such as chronic pulmonary disease
* Patients with asthma
* Patients with bradyarrhythmia
* Patients with concurrent liver and/or kidney dysfunction according to the latest laboratory test values within 14 days before the start of the pre-treatment observation period
* Patients with organic brain disorder such as elevated intracranial pressure, disturbance of consciousness/coma, or brain tumor
* Patients with any psychoneurologic complication and judged incapable of self assessment
* Patients with a history of drug dependency or narcotic abuse
* Patients with a history of hypersensitivity to fentanyl or any other opioid analgesic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2004-12; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Patient's global assessments of pain

SECONDARY OUTCOMES:
Physician's global assessments, pain intensity (Visual Analog Scale: VAS), pain intensity (categorical scale), total pain duration per day, and dose of rescue medication, Adverse events, laboratory values, and vital signs. Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.